CLINICAL TRIAL: NCT04303949
Title: Apply Gender Perspective Based Multi-media E-book to Enhance the Care Quality of a Second-Trimester Termination Due to Fetal Anomaly：for Parents and Nursing Professionals
Brief Title: Multi-Media E-Book for Second-Trimester Termination Due to Fetal Anomaly
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: CMUH108-REC1-077
Record Dates: First submitted 2019-12-03; First posted 2020-03-11 (Actual); Last update posted 2020-03-11 (Actual); Status verified 2020-03

CONDITIONS: Termination of Pregnancy
Keywords: Termination; Fetal anomaly; Gender; Grief; Nursing; e-book
MeSH Terms: conditions — Congenital Abnormalities; Coitus

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): e-book for termination
  Interventions: Other: Behavioral:
- Control (Other): routine care Written form health education
  Interventions: Other: Behavioral:

INTERVENTIONS:
Other: Behavioral: — Facilitating couples reduce anxiety, depression and grief through e-book education.

SUMMARY:
The subjects of this study are married couples who received termination of pregnancy, the main purpose is to explore the effectiveness of the e-book education model. Outcome indicators include anxiety, depression, and grief, as well as the satisfaction of the education.

DETAILED DESCRIPTION:
1. Study design: The study subjects were couples of obstetric inpatients who would receive termination of pregnancy. Both groups were assessed by the obstetrician in the outpatient clinic who must be admitted to the hospital to terminate the pregnancy. After receiving consent, a pre-test is performed in the clinic. The pre-test included questionnaires (basic attribute, State-Trait Anxiety Inventory (STAI) - the State Anxiety Scale (S-Anxiety), Perinatal Grief Scale (PGS), Beck Depression Inventory). After complete pre-teat, study nurse will provide the experimental group a QR Code to enter the cloud system (Hama Star e-book network platform), enable the couples to read the content at home; the control group receives traditional oral instructions. When the experimental group entered the delivery room, the researcher used the Hama Star e-book network platform to play the content of the termination of pregnancy e-book education model, and discussed the content with them; the control group receives regular traditional education model, with booklet and oral instructions, the intervention is about 20-25 minutes. The experimental group is able to use e-books as needed during induction, hospitalization, and after discharge. Two post-tests are conducted for follow-up. Both groups write the first post-test questionnaire (State-Trait Anxiety Inventory (STAI) - the State Anxiety Scale (S-Anxiety), Perinatal Grief Scale (PGS), Beck Depression Inventory) 60 minutes after education. Then, complete the second post-test questionnaire at the next appointment a month after.
2. Randomization Process: This study used a two-group pre- and post-test mode in experimental design, and random allocation to assign subjects into experimental and control groups. Participants were randomly allocated to the experimental or control group in a 1:1 ratio using the network randomization tool (www.randomizer.org/).
3. Sample size calculation:G-power version 3.1 was used to calculate the required sample size for the study. Set power 0.8, α = 0.05, based on the effectiveness (effect 0.30), the number of samples required for each group in this study is 32, because the tracking period is up to half a year, with a loss rate 50%, the two groups need a total of 96 participants.

ELIGIBILITY:
Inclusion Criteria:

1. At least 20 years old
2. Consciousness clear and capable of complete the questionnaires
3. Able to communicate in Mandarin or Taiwanese
4. Agree to participate in the study and sign the consent

Exclusion Criteria:

1. Emergency admissions for induction.
2. Non-medical reasons and pay own expenses to terminate the pregnancy
3. Have psychiatric illness history or other disorders that affect cognitive function

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2020-03-20 (Estimated); Primary Completion 2021-07-30 (Estimated); Study Completion 2021-07-30 (Estimated)

PRIMARY OUTCOMES:
Change in Anxiety level | The experimental group and the control group will accept the pretest and post-test before intervention, take another test after one month.
  State-Trait Anxiety Inventory State Anxiety (STAI-S) is used to measure the anxiety levels. State Anxiety refers to a temporary emotional state that changes over time, including the subjective perception of tension, anxiety, and fear. A total of 20 questions, the higher the score, the higher the degree of anxiety, the lower the score, the lighter the degree of anxiety. 20 - 39 means mild anxiety; 40 - 59 means moderate anxiety; 60 - 80 means severe anxiety. This scale has been widely used for many years to measure the anxiety of various conditions and has good reliability and validity.
Change in Grief Level | The experimental group and the control group will accept the pretest and post-test before intervention, take another test after six months.
  This study used the Perinatal Grief Scale (PGS) (1989) as a tool to measure the degree of a grief response, and Cronbach α value is 0.95. The questionnaire includes three aspects of Active Grief, Difficulty Coping and Despair, each aspect has 11 questions, a total of 33 questions. The total amount is calculated by the degree of sadness, from "very agree" to 1 point, "disagree" to 2 points, "not agreeing or denying" 3 Points, "Agree" 4 points, "very agree" 5 points, the total score is 33-165 points, the higher the score, the higher the level of sadness. It can be used as a measurement for predicting subjects with long-term grief.
Change in Depression Level | The experimental group and the control group will accept the pretest and post-test before intervention, take another test after six months.
  Beck Depression Inventory (BDI-II) is used to measure the level of depression. The content of the scale contains a total of 21 questions, each of which has four options according to the severity level, and scores ranging from 0 to 3 points.
Learning Motivational Change | The experimental group and the control group will accept the pretest and post-test before intervention, take another test after six months.
  Include learning motivation of sexual harassment Contains the learner's attention to the teaching material (12 questions), relevance (9 questions), confidence (9 questions), satisfaction (6 questions) and other learning motivation, a total of 36 questions, use Likert five-point scale, scoring method from 5 (very agreeable) to 1 (very disagree), the score range from 36-180 points, the higher the total score of the scale, the stronger the motivation of learning.

CONTACTS AND LOCATIONS:
Overall Officials: Ya-Ling Tzeng, PhD, Principal Investigator — China Medical University, Taiwan